CLINICAL TRIAL: NCT00365599
Title: Phase II Trial of Suberoylanilide Hydroxamic Acid (SAHA, Vorinostat) in Combination With Tamoxifen for Patients With Advanced Breast Cancer Who Have Failed Prior Anti-hormonal Therapy.
Brief Title: Phase II Trial of SAHA & Tamoxifen for Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-14662
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Suberoylanilide hydroxamic acid (SAHA); Vorinostat; Tamoxifen; Anti-hormonal therapy; Estrogen receptor positive; Progesterone receptor positive; Metastatic disease; Aromatase inhibitors (Ais); Histone deacetylase (HDAC) inhibitors; Selective estrogen receptor modulators(SERMS)
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Bulbo-Spinal Atrophy, X-Linked | interventions — Vorinostat; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vorinostat and Tamoxifen (Experimental): As outlined in Intervention descriptions
  Interventions: Drug: suberoylanilide hydroxamic acid (SAHA, Vorinostat); Drug: tamoxifen citrate (Tamoxifen)

INTERVENTIONS:
Drug: suberoylanilide hydroxamic acid (SAHA, Vorinostat) — Vorinostat will be used to potentiate the effects of tamoxifen or overcome tamoxifen resistance. All patients will receive vorinostat at 400 mg by mouth (po) daily for 3 out of 4 weeks. Responses will be assessed after 2 cycles (8 weeks + 4 days).
  Other Names: SAHA; Vorinostat; NSC #701852
Drug: tamoxifen citrate (Tamoxifen) — Tamoxifen will be given once daily at 20 mg. Tamoxifen will be given continuously. Responses will be assessed after 2 cycles (8 weeks + 4 days).
  Other Names: Nolvadex; Tam; Tamoxifen

SUMMARY:
Phase II trial to explore the efficacy of vorinostat and tamoxifen combined.

DETAILED DESCRIPTION:
Phase II trial to explore the efficacy of vorinostat and tamoxifen combined. Tamoxifen will be given once daily, continuously. Vorinostat will be given daily for 3 out of 4 weeks (a cycle). Responses will be assessed (restaged) after 2 cycles and toxicities will be captured continuously. Eligible patients will receive treatment in consecutive 4-week cycles, until progression of disease or unacceptable toxicity. Patients will be followed for evaluation of safety for at least 30 days after the last dose of the study drug.

Tests will be obtained pre-and post vorinostat treatment and correlated with plasma levels of vorinostat at the time of tumor biopsy and vorinostat doses; the tests will consist of:

* Patient history
* Physical exam (including height and weight)
* Toxicity assessment
* Pharmacokinetic (PK) sample
* Tumor fine needle aspirate (FNA)
* Peripheral Blood Mononuclear Cells (PBMC)
* Standard labs and Chemistry Profile
* Carcinoembryonic antigen (CEA), cancer antigen (Ca) 15-3, Ca 125 (If clinically indicated)
* Pregnancy Test
* Computed tomography (CT) scans, and magnetic resonance imaging (MRI)

Documentation of response and progression will be evaluated in this study using the Response Evaluation Criteria in Solid Tumors (RECIST).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have cytologically/histologically documented locally advanced or metastatic breast cancer with either:

  1. Progression on treatment with any aromatase inhibitor for metastatic disease;
  2. Recurrence while on adjuvant aromatase inhibitors or within 12 months of completion;
  3. Recurrence after having completed adjuvant tamoxifen for at least 12 months;
  4. Patient who are not candidates for or are intolerant of aromatase inhibitor treatment;
  5. Patients are allowed (but not required) to have one prior chemotherapy regimen for metastatic disease.
* Tumors must express estrogen or progesterone receptor.
* Patients are eligible regardless of the menopausal status.
* Age > 18 years old
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Patients must be able to give informed consent and able to follow guidelines given in the study.
* Patients must have acceptable organ function, as defined by the following laboratory parameters: white blood count (WBC) >3.0 x 10^9/L; absolute neutrophil count (ANC) >1.5 x 10^9/L; hemoglobin (Hgb) >10.0g/dL; platelets (PLT) >100 x 10^9/L, Bilirubin < 2.0 mg/dl, aspartate aminotransferase/alanine aminotransferase (AST/ALT) < 2.5 X upper limit of normal (ULN), Creatinine <1.8 mg/dl (Creatinine clearance >60 ml/min).
* Women of childbearing age must have a negative pregnancy test. All patients of reproductive potential must use an effective method of contraception during the study and 6 months following termination of treatment. (Not applicable to patients with bilateral oophorectomy and/or hysterectomy or to female patients who are older than 50 years and have not had a menstrual cycle in more than one year.
* Patients must have measurable disease by RECIST criteria by staging studies performed within 30 days of enrollment. For patients with bone only disease: For this protocol isolated bone lesions can be classified as target lesions if they are measurable by MRI at screening and must be followed by MRI.
* Both men and women of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Patients must not have received tamoxifen for metastatic disease.
* Patients must not have evidence of significant active infection (e.g., pneumonia, cellulitis, wound abscess, etc.) at time of study entry.
* Patients must be disease-free of prior invasive malignancies for > 5 years with the exception of: curatively-treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix.
* Pregnant and breast-feeding women are excluded from the study because effects on the fetus are unknown and there may be a risk of increased fetal wastage.
* Patients with uncontrolled central nervous system (CNS) metastasis or a history of seizures are excluded. Patients with stable CNS metastasis (either surgically resected, treated with gamma knife or stable for 3 months following whole brain radiation therapy [WBRT] are eligible). Patients with stable brain metastases will need an MRI within 4 weeks prior to start of therapy.
* Patients may not be receiving any other investigational agents and must have stopped all other histone deacetylase inhibitors (including Valproic acid) or other hormonal therapies.
* Patients must have discontinued their prior therapies for breast cancer and radiation therapy for a minimum of 3 weeks, patient is excluded if radiation therapy was given to a single measurable lesion and the disease is otherwise not measurable.
* Patients are excluded if they have any known hypersensitivity reaction to tamoxifen.
* Patient with a history of blood clots are not eligible.
* Women who have abnormal vaginal bleeding and/or endometrial hyperplasia or cancer are not eligible.
* Patients with evidence of visceral crisis are not eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-02; Primary Completion 2011-04 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Minton, D.O., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (8):
- United States (8):
  - University of California, San Francisco, California
  - Bethesda Memorial Hospital Research Center, Boynton Beach, Florida
  - M.D. Anderson of Orlando, Orlando, Florida
  - Fawcett Memorial Hospital, Port Charlotte, Florida
  - Martin Memorial Cancer Center, Stuart, Florida
  - Tallahassee Memorial HealthCare, Inc., Tallahassee, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - St. Joseph's/Candler, Savannah, Georgia

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials Website — http://www.moffitt.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Estrogen or progesterone receptor positive advanced breast cancer: Postmenopausal, failed first-line therapy with aromatase inhibitor or recurred within 12 months of adjuvant treatments with aromatase inhibitors; Premenopausal, recurred >12 months after adjuvant tamoxifen or never treated with tamoxifen; Not candidate for aromatase inhibitor
Groups:
- Vorinostat and Tamoxifen: Vorinostat and Tamoxifen as outlined in Intervention Descriptions
Period: Overall Study
Arm/Group | Vorinostat and Tamoxifen
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vorinostat and Tamoxifen
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 6
Age, Customized [Median (Full Range); unit: years] | 56 [33 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response (OR)
Description: The Objective Response Rate. Response and progression were evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST). Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria. For the purposes of this study, patients were evaluated for response every 8 weeks. In addition to a baseline scan, confirmatory scans were also obtained ≥ 4 weeks following initial documentation of objective response.
Time Frame: 24 weeks
Population: All participants
Measure: Number; unit: participants
Arm/Group | Vorinostat and Tamoxifen
Number analyzed (Participants) | 43
participants | 8

2. Secondary Outcome: Time to Progression (TTP)
Description: The median response duration in months. Response and progression were evaluated in this study using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: Up to 30 months
Population: All participants
Measure: Median (Full Range); unit: months
Arm/Group | Vorinostat and Tamoxifen
Number analyzed (Participants) | 43
months | 10.3 [8.1 to 12.4]

3. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Safety evaluation according to descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.
Time Frame: 4 years, 7 months
Population: All participants
Measure: Number; unit: participants
Arm/Group | Vorinostat and Tamoxifen
Number analyzed (Participants) | 43
participants | 4

ADVERSE EVENTS:
Time Frame: 4 years, 7 months
Arm/Group | Vorinostat and Tamoxifen
Serious Adverse Events (participants affected / at risk) | 4/43
Other Adverse Events (participants affected / at risk) | 33/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat and Tamoxifen (N=43)
Anorexia (Gastrointestinal disorders) | 1 (1) — Grade 2, probably related
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) — Grade 3, possibly related
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 1 (1) — Grade 2, possibly related
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) — Grade 3, related
Platelets (Blood and lymphatic system disorders) | 1 (1) — Grade 4, related
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1) — Grade 3, possibly related
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2) — Grade 4, possibly related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat and Tamoxifen (N=43)
Alopecia - Grade 2 (Skin and subcutaneous tissue disorders) | 4 (4)
Anorexia/weight loss - Grade 2 (Gastrointestinal disorders) | 7 (11)
Anorexia/weight loss - Grade 3 (Gastrointestinal disorders) | 4 (4)
Deep vein thrombosis/pulmonary embolish (DVT/PE) - Grade 4 (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Diarrhea - Grade 2 (Gastrointestinal disorders) | 7 (8) — (There was also one Grade 3 event, below the Frequency Threshold for reporting)
Fatigue - Grade 2 (General disorders) | 8 (16)
Fatigue - Grade 3 (General disorders) | 7 (8)
Hepatic dysfunction (alanine aminotransferase/aspartate aminotransferase [ALT/AST]) - Grade 2 (Metabolism and nutrition disorders) | 3 (8) — (There was also one Grade 3 event, below the Frequency Threshold for reporting)
Hyperglycemia - Grade 2 (Metabolism and nutrition disorders) | 5 (11) — (There were also 2 Grade 3 events, below the Frequency Threshold for reporting)
Leukopenia - Grade 2 (Blood and lymphatic system disorders) | 4 (9) — (There were also 2 Grade 3 events, below the Frequency Threshold for reporting)
Lymphopenia - Grade 2 (Blood and lymphatic system disorders) | 5 (16)
Lymphopenia - Grade 3 (Blood and lymphatic system disorders) | 6 (6)
Nausea - Grade 2 (Gastrointestinal disorders) | 8 (13)
Neutropenia - Grade 2 (Blood and lymphatic system disorders) | 5 (5)
Neutropenia - Grade 3 (Blood and lymphatic system disorders) | 7 (7)
Thrombocytopenia - Grade 2 (Blood and lymphatic system disorders) | 4 (7)
Thrombocytopenia - Grade 3 (Blood and lymphatic system disorders) | 3 (3) — (There was also one Grade 4 event, below the Frequency Threshold for reporting)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No